CLINICAL TRIAL: NCT06122623
Title: Education Program for Enhancing Healthcare Students' Attitudes Toward People Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Collaborators: Tokyo University (Other); Kawasaki City College of Nursing (Unknown)
Responsible Party: Principal Investigator, Dianis Wulan Sari, Principal Investigator, Universitas Airlangga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UAirlangga
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Dementia
Keywords: Aged; Dementia; Healthcare student; Education program; Long-term care
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-arm pre-post approach will be employed in this study; (Other): There will be no control group. All participants will receive the same treatment. The intervention to be used will be a gaming education program conducted once with each participant.
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Health Education — As previously mentioned, the intervention for this study will be a gaming education program that will be conducted once with each participant. Implementation of the program will occur at different times. Each performance will include a maximum of 60 participants who will be divided into small groups within the same room. Seven to 10 participants will comprise a small group, and each group will have one facilitator. The facilitator will be either a member of the research team or a Health lecturer who will be recruited and trained by the Japanese and Indonesian research teams.

SUMMARY:
The aim of this single-arm pre-post study is to examine the effectiveness of gaming-based dementia educational programs for enhancing healthcare students' attitudes toward people living with dementia (PLWD). The main questions we intend to answer follow:

* What are the attitudes toward PLWD, intentions to help PLWD, knowledge of dementia, and stigma of PLWD before and after participation in the gaming-based dementia education program?
* What is the effect of gaming-based dementia education programs on enhancing attitudes toward PLWD?

Participants will volunteer for the class education program, which will last about 90 minutes. Participants can attend the class only once. This education program based on gaming tools will be structured with a lecture on dementia, N-impro (gaming tools), and bad/good short dramas. The gaming education program will be included in dementia-related courses.

DETAILED DESCRIPTION:
Participants in this study will be healthcare students at an Indonesian university (i.e., nursing students, public health students, etc.) enrolled in the semesters and courses designated for implementation of this educational program. For example, nursing students at Airlangga University will be among students in their fifth semester. Prospective participants will be given new ID numbers to ensure that their student ID numbers are undetected. The protocol for this study was reviewed and approved by an ethical committee of the Faculty of Nursing at Airlangga University.

Regarding recruitment, all candidate participants will be identified from the university's e-learning portal data. Students registered in the courses selected for implementation of this education program will have their data recorded at the beginning of the odd semester for the 2023/2024 academic year. Potentially eligible candidates will receive comprehensive study information and an invitation to participate.

The courses coordinator and Principal Investigator (PI) will explain the Semester Learning Plan and curriculum for the selected courses at the beginning of the semester. An overview of the research session's implementation will be presented, while detailed research procedures will be explained shortly before research is undertaken. An announcement regarding implementation of the research will be made approximately one week in advance, and recruitment will be carried out through Google Forms. Candidate participants will receive new IDs for this study and information about the schedule and location of the educational program through a class announcement three days prior.

On the intervention date, candidate participants will be present at the designated location and sign an attendance sheet using their new IDs. The PI will explain all stages of the study and reiterate regarding participants' freedom to withdraw at any time. The recruitment of study participants will not involve coercion. Students who choose not to participate in this study will still receive regular dementia-related materials through the university's e-learning portal, but they will not receive the game-based education program. Students who agree to participate in the study will provide informed consent. Further, participants in the educational program will complete a questionnaire before and after its implementation.

ELIGIBILITY:
Inclusion Criteria:

Healthcare students enrolled in the designated semester and courses that align with the program's implementation

Exclusion Criteria: -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Attitude toward people living with dementia | Time Frame: 5-7 minutes for completion of the questionnaire
  We will examine participants' attitudes toward people living with dementia with the Attitudes Toward People with Dementia Scale (Kim K, Kuroda K. Factors related to attitudes toward people with dementia development attitude toward dementia scale and dementia knowledge scale. Bulletin of Social Medicine. 2011; 28 (1), 43-55). The original study was published in Japanese. We performed forward-backwards translation to produce the Indonesian language version.
  The total number of items in the questionnaire is 14. This scale has a 4-point Linkert scale ranging from 1 (disagree) to 4 (agree). There consists of four subscales: tolerance (five items), refusal (four items), feeling of distance (three items), and affinity 8two items). The total score ranged from 14 to 56, with a higher score indicating a more favourable attitude.

SECONDARY OUTCOMES:
Knowledge of dementia | Time Frame: 5-7 minutes
  Knowledge of dementia will be measured using 15 items of the Dementia-Related Knowledge Scale developed by (Kim & Kuroda, 2011), which assesses the knowledge of dementia, symptoms, treatments, and diagnosis of dementia. This dementia knowledge scale will ask respondents to answer with a 4-point Likert scale from disagree to agree. The author will calculate the total score of knowledge of dementia. The total score ranged from 15 to 60, with a higher score indicating a higher knowledge of dementia.
Intention for helping behaviors toward people living with dementia | Time Frame: 2-3 minutes
  To assess the Intention for helping behaviours toward people living with dementia, intended helping behaviours will be measured using four vignettes based on a previous study by Matsumoto et al. (2022). The vignettes describe situations in which people living with dementia may need assistance. Intended helping behaviours will be measured using a 4-point Likert scale (1= strongly disagree, 2= disagree, 3= agree, and 4= strongly agree). The higher score indicates a higher intention of helping behaviours people living with dementia.
Fraboni's Scale of Ageism (FSA) | Time Frame: 5-7 minutes
  To assess ageism associated with people living with dementia, we will use the Fraboni Scale of Ageism (FSA) short version of 19 items. The FSA short version consists of 19 items. That rate the negative opinion towards older people using the Likert scale (1= strongly disagree, 2= disagree, 3= agree, and 4= strongly agree). Statements representing positive rather than negative opinions towards older adults had reversed scoring (item numbers 13-16). Possible scores of FSA ranged from 19-76. The higher score indicates a higher level of ageism.

CONTACTS AND LOCATIONS:
Overall Officials: Dianis Wulan Sari, Ph.D, Principal Investigator — Universitas Airlangga
Locations (1):
- Universitas Airlangga, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The IPD associated with participants' real IDs will be retained only by the PI of this study.
  New datasets will use new IDs so that only the PI can link the research data to participants' original IDs.
  Datasets that use the new IDs will be shared with the research team for data processing purposes (statistical analysis plan, SAP) and publication. All data will be stored for five years (November 2023-November 2028).
  Datasets will not be made public and will only be shared with the project's research team.

REFERENCES:
- [Background] Fraboni, M., Saltstone, R., & Hughes, S. (1990). The Fraboni Scale of Ageism (FSA): An Attempt at a More Precise Measure of Ageism. Canadian Journal on Aging / La Revue Canadienne Du Vieillissement, 9(1), 56-66.
- [Background] Lane AP, Yu FCH. Person-centered attitudes mediate the association between dementia knowledge and help-giving intentions in Singapore. Int Psychogeriatr. 2020 Mar;32(3):413-414. doi: 10.1017/S1041610219000796. No abstract available. PMID 31309909
- [Result] Blay SL, Toledo Pisa Peluso E. Public stigma: the community's tolerance of Alzheimer disease. Am J Geriatr Psychiatry. 2010 Feb;18(2):163-71. doi: 10.1097/JGP.0b013e3181bea900. PMID 20104072
- [Result] Brannelly T. Sustaining citizenship: people with dementia and the phenomenon of social death. Nurs Ethics. 2011 Sep;18(5):662-71. doi: 10.1177/0969733011408049. PMID 21893577
- [Result] Harada, K., Sugisawa, H., Shibata, H., Yamada, Y., & Sugihara, Y. (2004). Measurement and Correlates of Ageism Among Japanese Young Men Living in Urban Areas. The Gerontologist, 44(Special_Issue_I), 1-672.
- [Result] Kim, K., & Kuroda, K. (2011). Factors related to attitudes toward people with dementia: Development Attitude Toward Dementia Scale and Dementia Knowledge Scale. Bulletin of Social Medicine, 28(1), 43-56 (in Japanese).
- [Result] Malta S, Doyle C. Butler's three constructs of ageism in Australasian Journal on Ageing [corrected]. Australas J Ageing. 2016 Dec;35(4):232-235. doi: 10.1111/ajag.12363. No abstract available. PMID 27933747
- [Result] Matsumoto H, Igarashi A, Sakka M, Takaoka M, Kugai H, Ito K, Yamamoto-Mitani N. A Two-Step Model for Encouraging the General Public to Exhibit Helping Behaviors Toward People Living With Dementia. Innov Aging. 2022 Apr 14;6(3):igac023. doi: 10.1093/geroni/igac023. eCollection 2022. PMID 35663276
- [Result] Stites SD, Milne R, Karlawish J. Advances in Alzheimer's imaging are changing the experience of Alzheimer's disease. Alzheimers Dement (Amst). 2018 Mar 19;10:285-300. doi: 10.1016/j.dadm.2018.02.006. eCollection 2018. PMID 29780873
- [Derived] Sari DW, Kugai H, Igarashi A, Takaoka M, Matsumoto H, Suzuki H, Wu J, Fitryasari R, Nasifah IA, Has EMM, Yamamoto-Mitani N. Education Program for Enhancing Health Care Students' Attitudes Toward People Living With Dementia: Protocol for a Single-Arm Pre-Post Study. JMIR Res Protoc. 2024 Sep 18;13:e62654. doi: 10.2196/62654. PMID 39293050